CLINICAL TRIAL: NCT06908174
Title: Differences in Prosocial Behaviors and Related Brain Networks in Children With Autism and Typical Development
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: ShanghaiTech University (Other)
Responsible Party: Sponsor
Other Study IDs: brainpro2022-cross-sectional
Record Dates: First submitted 2025-02-19; First posted 2025-04-03 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Healthy
Keywords: autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case group: Subjects in the case group are diagnosed with autism spectrum disorder according to DSM-V and clinical observation.
  Interventions: Diagnostic Test: ADOS-2
- Control group: Subjects in the control group are healthy children without serious chronic or congenital diseases.

INTERVENTIONS:
Diagnostic Test: ADOS-2 — The subjects in case group will receive the ADOS-2 assessment to confirm their diagnosis.
  Groups: Case group

SUMMARY:
The goal of this observational study is to compare the brain functional network between children with autism and typical development, using magnetic resonance imaging (MRI), electroencephalogram/event-related potentials(EEG/ERPs) and functional Near Infrared Spectrum(fNIRs). The main questions it aims to answer are as follows: 1. What are the differences of the functional brain network between autism and TD children? 2. What are the differences of the brain activity in response to special social stimulus between autism and TD children? Participants will receive developmental/intelligence assessments (Griffiths Mental Developmental Scales/Wechsler Preschool and Primary Scale of Intelligence-IV/Wechsler Intelligence Scale for Children-IV for children of different ages), social assessments(Autism Diagnostic Observation Schedule-2nd Edition/Social Communication Questionnaire), EEG/ERPs and fNIRs in resting and task states, and head MRI in natural sleeping state(without sedative).

DETAILED DESCRIPTION:
The cross-sectional observational study will be performed to compare the differences of functional brain network and reactions to social stimulus between children with autism and typical development. The investigators will recruit children aged between 2 to 17 years and 11 months old. They need to receive the mentioned assessments and medical examinations for at least once.

ELIGIBILITY:
Case group:

Inclusion Criteria:

1. Children diagnosed with ASD according to a clinical judgement based on the criteria of ASD in DSM-5 and further confirmed with ADOS-2;
2. Ages 2-17 years;
3. Parents/caregivers understand the content of the study and agree to participate in.

Exclusion Criteria:

1. Rett Syndrome, Fragile X Syndrome, Angelman Syndrome, Prader-Willi Syndrome, tuberous sclerosis, and other syndromes caused by known genetic defects or inherited metabolic diseases;
2. Children with brain injuries, specific chronic or congenital diseases.
3. The gestational age is less than 37 weeks, or the birth weight is lower than 2500g.
4. Children cannot receive the head MRI examination.

Control group:

Inclusion Criteria:

1. Healthy children age between 2 to 17 years.
2. Children without the family history of ASD or other neurodevelopmental/mental diseases.
3. Parents/caregivers understand the content of the study and agree to participate in.

Exclusion Criteria:

1. Children with brain injuries, specific chronic or congenital diseases.
2. The gestational age is less than 37 weeks, or the birth weight is lower than 2500g.
3. Children cannot receive the head MRI examination.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The observation study will be performed in children with ASD and healthy, typically developing children.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
clinical diagnosis | Baseline (during 2 to 17 years old).
  Clinicians will diagnose subjects as ASD, other neurodevelopmental disorders, or typical developing children, using DSM-5 and ADOS-2. The minimum and maximum scores of ADOS-2 are 0 and 28, and the comparison score of ADOS-2 ranges from 1 to 10, in which higher scores mean a worse outcome.
Latencies in event related potentials(ERPs) | Baseline (during 2 to 17 years old).
  The investigators will explore the differences of N1/N2, P3/LPP and N400 in event related potentials (ERPs) between case and control groups (children with ASD and typical development) in responses to special prosocial stimulus, and also in false belief tasks. Event related potentials (ERPs) will be tested using eego™ mylab of ANT Neuro company.
Amplitudes in ERPs | Baseline (during 2 to 17 years old).
  Amplitudes of N1/N2, P3/LPP and N400 will be compared between children with autism spectrum disorder and typical development.
nuclear magnetic resonance imaging(MRI) | Baseline (during 2 to 17 years old).
  Cranial MRI data, including sMRI and fMRI, will be collected during subjects are in natural asleep or awake, using uMR 890 3T of United Imaging company.
Changes in the concentrations of Oxygenated Hemoglobin (HbO) and deoxygenated Hemoglobin (HbR) during interactions | Baseline (during 2 to 17 years old).
  The investigators will explore inter-group differences of children with ASD and typical development in the concentrations of HbO and HbR during social communication scenes between participants and investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Xu, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No